CLINICAL TRIAL: NCT04587180
Title: The Correlation Between the Bone Mineral Density of the Proximal Humerus and Cutting-through at the Greater Tuberosity in Arthroscopic Suture-bridge Rotator Cuff Repair
Brief Title: Cutting-through at the Greater Tuberosity
Status: Completed | Type: Observational
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Collaborators: Hallym University (Other)
Responsible Party: Principal Investigator, Jung-Taek Hwang, Associate Professor, Chuncheon Sacred Heart Hospital
Other Study IDs: 2014-33
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Rotator Cuff Tears
Keywords: rotator cuff tear; cutting-through; Bone mineral density; suture-bridge repair
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patients with cutting-through: Patients who had cutting-through during the lateral knotless anchor fixation.
  Interventions: Procedure: Arthroscopic suture-bridge rotator cuff repair
- Patients without cutting-through: Patients who didn't have cutting-through during the lateral knotless anchor fixation.
  Interventions: Procedure: Arthroscopic suture-bridge rotator cuff repair

INTERVENTIONS:
Procedure: Arthroscopic suture-bridge rotator cuff repair — Arthroscopic suture-bridge repair is a widely used and universal surgical method for symptomatic rotator cuff tear patients. It is arthroscopic surgery to reattach ruptured rotator cuff tendons to the original insertion (greater tuberosity) using medial and lateral row anchors.

SUMMARY:
The investigators evaluated the correlation between cutting-through at the greater tuberosity (GT) just medial to the lateral knotless anchor in arthroscopic suture-bridge rotator cuff repair and the bone mineral density (BMD) of the lumbar spine, hip and GT of the proximal humerus and to evaluate factors and clinical outcomes related to cutting-through at the GT.

DETAILED DESCRIPTION:
Seventy-eight patients who underwent arthroscopic suture-bridge rotator cuff repair and who had undergone dual energy X-ray absorptiometry (DEXA) scans before surgery were included. Patients were divided into two groups: patients who had cutting-through (46, group I) and patients who did not (32, group II). Clinical and radiological data including demographics, BMDs, fatty infiltration of rotator cuff muscles, tear size, tear involvement, VAS pain score, and ASES score were analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Primary arthroscopic repair for a symptomatic full-thickness rotator cuff tear identified by preoperative MRI
2. Dual energy X-ray absorptiometry (DEXA) to evaluate the BMD of the lumbar spine and hip, as a standardized measurement, and the GT of the affected proximal humerus
3. Follow up for a minimum of 2 years after the primary surgery.

Exclusion Criteria:

1. Primary arthroscopic repair due to partial-thickness rotator cuff tear or an isolated subscapularis tear
2. Primary suture-bridge repair with 3 or more lateral-knotless anchors
3. Previous history of fractures or surgeries on the affected shoulder
4. Shoulder instability
5. Glenohumeral osteoarthritis
6. Neurologic or systemic disease diseases influencing the shoulder joint 7 History of infection of the shoulder joint

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with arthroscopic rotator cuff suture-bridge repair for full-thickness rotator cuff tears
Sampling Method: Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2015-10-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
The occurrence of cutting-through | During the surgery
  The occurrence of cortical breakage of the GT just medial to the lateral knotless anchor hole due to the tension of the sutures from the medial anchor
Visual Analog Scale (VAS) Pain Score | 2 years after surgery
  The VAS pain score was based on a scale from 0 to 10, where 0 indicated no pain and 10 indicated severe pain
American Shoulder and Elbow Surgeons (ASES) score | 2 years after surgery
  American Shoulder and Elbow Surgeons score for estimating shoulder function was based on a score from 0 to 100, where 0 indicated poor outcome and 100 indicated excellent outcome.
Greater tuberosity bone mineral density | preoperatively
  GT BMD was measured using the predefined region of interest (ROI). Dividing the humeral head into three columns of even width, we defined a 1x1-cm2-sized square in the center of the lateral column as ROI.
Lumbar spine bone mineral density | preoperatively
  Measured by using standard techniques according to the manufacturer and the International Society for Clinical Densitometry guidelines.
Hip bone mineral density | preoperatively
  Measured by using standard techniques according to the manufacturer and the International Society for Clinical Densitometry guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Taek Hwang, MD, PhD, Principal Investigator — Chuncheon Sacred Heart Hospital

REFERENCES:
- [Background] Oh JH, Song BW, Lee YS. Measurement of volumetric bone mineral density in proximal humerus using quantitative computed tomography in patients with unilateral rotator cuff tear. J Shoulder Elbow Surg. 2014 Jul;23(7):993-1002. doi: 10.1016/j.jse.2013.09.024. Epub 2013 Dec 31. PMID 24388151
- [Background] Oh JH, Song BW, Kim SH, Choi JA, Lee JW, Chung SW, Rhie TY. The measurement of bone mineral density of bilateral proximal humeri using DXA in patients with unilateral rotator cuff tear. Osteoporos Int. 2014 Nov;25(11):2639-48. doi: 10.1007/s00198-014-2795-1. Epub 2014 Jul 16. PMID 25027108
- [Background] Pogorzelski J, Fritz EM, Horan MP, Katthagen JC, Hussain ZB, Godin JA, Millett PJ. Minimum Five-year Outcomes and Clinical Survivorship for Arthroscopic Transosseous-equivalent Double-row Rotator Cuff Repair. J Am Acad Orthop Surg. 2019 Dec 15;27(24):e1093-e1101. doi: 10.5435/JAAOS-D-18-00519. PMID 31805019
- [Background] Ono Y, Woodmass JM, Nelson AA, Boorman RS, Thornton GM, Lo IK. Knotless anchors with sutures external to the anchor body may be at risk for suture cutting through osteopenic bone. Bone Joint Res. 2016 Jun;5(6):269-75. doi: 10.1302/2046-3758.56.2000535. PMID 27357383
- [Derived] Lee S, Hwang JT, Lee SS, Lee JH, Kim TY. Greater Tuberosity Bone Mineral Density and Rotator Cuff Tear Size Are Independent Factors Associated With Cutting-Through in Arthroscopic Suture-Bridge Rotator Cuff Repair. Arthroscopy. 2021 Jul;37(7):2077-2086. doi: 10.1016/j.arthro.2021.01.059. Epub 2021 Feb 10. PMID 33581302